CLINICAL TRIAL: NCT03493425
Title: Phase II Randomized Trial of Neo-Adjuvant Chemotherapy Followed by Surgery and Post-Operative Radiation Versus Surgery and Post-Operative Radiation for Organ Preservation of T3 and T4a Nasal and Paranasal Sinus Squamous Cell Carcinoma (NPNSCC)
Brief Title: Chemotherapy Before Surgery and Radiation Therapy or Surgery and Radiation Therapy Alone in Treating Patients With Nasal and Paranasal Sinus Cancer That Can Be Removed by Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA3163; NCI-2017-01364 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA3163 (Other: ECOG-ACRIN Cancer Research Group); EA3163 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-04-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stage III Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma AJCC v7
MeSH Terms: interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (surgery, IMRT, cisplatin, carboplatin) (Active Comparator): Patients undergo standard of care surgery. Beginning 4-6 weeks after surgery, patients undergo image guided IMRT QD for 5 fractions per week for 30 fractions. Patients with positive margins/positive ECS in lymph nodes undergo image guided IMRT QD for 5 fractions per week for 30 fractions and cisplatin IV over 1-2 hours or carboplatin IV over 30 minutes (for patients who are ineligible to receive cisplatin) weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery
- Arm B (docetaxel, cisplatin, carboplatin, surgery, IMRT) (Experimental): Patients receive docetaxel IV over 1 hour and cisplatin IV over 1-2 hours on day 1. Patients who are ineligible to receive cisplatin receive carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery no later than 6 weeks following the last dose of chemotherapy. Beginning 4-6 weeks after surgery, patients undergo image guided IMRT QD for 5 fractions per week for 30 fractions. Patients with positive margins/positive ECS in lymph nodes undergo image guided IMRT QD for 5 fractions per week for 30 fractions and cisplatin IV or carboplatin IV weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Docetaxel; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm B (docetaxel, cisplatin, carboplatin, surgery, IMRT)
Radiation: Image Guided Radiation Therapy — Undergo image guided IMRT
  Other Names: IGRT; image-guided radiation therapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo image guided IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery

SUMMARY:
This randomized phase II trial studies how well chemotherapy before surgery and radiation therapy works compared to surgery and radiation therapy alone in treating patients with nasal and paranasal sinus cancer that can be removed by surgery. Drugs used in chemotherapy, such as docetaxel, cisplatin, and carboplatin work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving chemotherapy before surgery and radiation therapy may make the tumor smaller and reduce the amount of normal tissue that needs to be removed and treated with radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the structure preservation rate for patients with locally advanced resectable nasal and paranasal sinus squamous cell carcinoma (NPNSCC) with or without neoadjuvant therapy; all patients will undergo surgical resection and postoperative standard care.

II. Evaluate overall survival (OS) for patients with locally advanced resectable NPNSCC with or without neoadjuvant therapy followed by surgical resection and postoperative standard care.

SECONDARY OBJECTIVES:

I. Evaluate progression-free survival (PFS) for this patient population. II. Examine the rate of structure preservation for the orbit (freedom from orbital exenteration).

III. Evaluate site reported p16 data and correlate with outcome. IV. Determine the accuracy of baseline/post-chemotherapy magnetic resonance imaging (MRI) and fludeoxyglucose F-18 positron emission tomography/computed tomography (FDG PET/CT)-based prediction of orbit and skull base preservation.

V. Determine the accuracy of baseline/post-chemotherapy MRI and/or FDG PET/CT-based prediction of 2-year overall survival.

TERTIARY OBJECTIVES:

I. To determine the effects of tobacco, operationalized as combustible tobacco (1a), other forms of tobacco (1b), and environmental tobacco exposure (ETS) (1c) on provider-reported cancer-treatment toxicity (adverse events [both clinical and hematologic] and dose modifications).

II. To determine the effects of tobacco on patient-reported physical symptoms and psychological symptoms.

III. To examine quitting behaviors and behavioral counseling/support and cessation medication utilization.

IV. To explore the effect of tobacco use and exposure on treatment duration, relative dose intensity, and therapeutic benefit.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo standard of care surgery. Beginning 4-6 weeks after surgery, patients undergo image guided intensity modulated radiation therapy (IMRT) once daily (QD) for 5 fractions per week for 30 fractions. Patients with positive margins/positive extracapsular spread (ECS) in lymph nodes undergo image guided IMRT QD for 5 fractions per week for 30 fractions and cisplatin intravenously (IV) over 1-2 hours or carboplatin IV over 30 minutes (for patients who are ineligible to receive cisplatin) weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive docetaxel IV over 1 hour and cisplatin IV over 1-2 hours on day 1. Patients who are ineligible to receive cisplatin receive carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery no later than 6 weeks following the last dose of chemotherapy. Beginning 4-6 weeks after surgery, patients undergo image guided IMRT QD for 5 fractions per week for 30 fractions. Patients with positive margins/positive ECS in lymph nodes undergo image guided IMRT QD for 5 fractions per week for 30 fractions and cisplatin IV over 1-2 hours or carboplatin IV over 30 minutes (for patients who are ineligible to receive cisplatin) weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if < 2 years from study entry and then every 6 months if 2-5 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* General physical condition compatible with the proposed chemotherapy and surgery
* Stage T3 or T4a, histologically-confirmed NPNSCC requiring orbital or skull base resection:

  * Stages T3 and T4a disease will be included regardless of nodal status (N0 or N1-3), provided that surgical therapy would require orbital or skull base resection
  * The surgical oncologist in each institution will determine the need for resection of the orbit OR base of skull at baseline for patients on both Arms A and B and following neo-adjuvant chemotherapy for patients on Arm B

    * Resection of skull base will be deemed necessary according to skull base bone erosion by CT or marrow involvement by MRI is noted; for any disease abutting the skull base; or for ethmoid sinus or frontal sinus involvement
    * Resection of orbital contents will be deemed necessary according to skull base society guidelines, based on involvement of periorbital fat documented by MRI imaging
* Patients must be deemed surgically resectable by the surgical teams at each institution and must have a determination of degree of anticipated structure preservation of orbit and skull base; this needs to be determined prior to randomization
* Patients may not be receiving investigational agents at time of registration, or at any time while on study and during the 4 weeks preceding enrollment
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel and/or both platinum-based chemotherapy agents are excluded; patient must be able to receive at least one of the two proposed chemotherapy regimens
* Patients with evidence of distant metastases or leptomeningeal disease (LMD) are excluded
* Patients must not have received previous irradiation for head and neck tumor, skull base, or brain tumors
* Patients with uncontrolled inter-current illnesses which in the opinion of the investigator will interfere with the ability to undergo therapy including chemotherapy are excluded
* Patients with a history of a different malignancy are excluded, unless the disease has not progressed for >= 2 years
* Absolute neutrophil count (ANC) > 1500/mm^3 =< 2 weeks prior to randomization
* Hemoglobin (Hgb) > 8.0 g/dL =< 2 weeks prior to randomization
* Platelet count > 100,000/mm^3 =< 2 weeks prior to randomization
* Creatinine clearance of > 60 ml/min; creatinine clearance may be measured or calculated; if calculating, creatinine clearance, use the Cockroft-Gault formula =< 2 weeks prior to randomization
* Total bilirubin within normal limits (must be obtained =< 2 weeks prior to randomization)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) must be within the range allowing for eligibility, must be obtained < 2 weeks prior to randomization
* Alkaline phosphatase must be within the range allowing for eligibility, must be obtained < 2 weeks prior to randomization
* Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated
* No current peripheral neuropathy > grade 2 at time of randomization
* Patients must not have any co-existing condition that would preclude full compliance with the study; no prior history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Women must not be pregnant or breast-feeding

  * All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study
* Patients must have measurable disease; MRI and/or PET/CT scans need to be performed within 2 weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Structure preservation rate defined as both skull base and orbit being preserved | Up to 5 years
  Fisher?s exact test will be used to compare the structure preservation rate between the two arms. The comparison between the two arms for structure preservation will be conducted separately (each at one-sided 0.05 significance level).
Overall survival (OS) | From date of randomization, censoring follow-up at last date of contact, assessed for up to 5 years
  Log rank test will be used to compare OS between the two arms. The comparison between the two arms for OS will be conducted separately (each at one-sided 0.05 significance level).

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Saba, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (140):
- United States (140):
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Adilbay D, Valero C, Fitzgerald C, Yuan A, Mimica X, Gupta P, Wong RJ, Shah JP, Patel SG, Ganly I, Cohen MA. Outcomes in surgical management of sinonasal malignancy-A single comprehensive cancer center experience. Head Neck. 2022 Apr;44(4):933-942. doi: 10.1002/hed.26989. Epub 2022 Jan 25. PMID 35080076